CLINICAL TRIAL: NCT06043960
Title: The Relationship Between Lower Limb Functionality, Foot Joint Position Sensation and Balance in Haemiplegic Patients
Status: Completed | Type: Observational
Sponsor: Karabuk University (Other)
Collaborators: Bolu Izzet Baysal Physiotherapy and Rehabilitation Training and Research Hospital (Unknown)
Responsible Party: Principal Investigator, Fatma Hale Altınkaya, INVESTIGATOR, Karabuk University
Other Study IDs: BAIBÜFTR
Record Dates: First submitted 2023-09-05; First posted 2023-09-21 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Being Between 40-80 Years Old; Being Diagnosed With Haemiplegia; Getting 20 Points or More in the Mini Mental Test; Volunteering to Participate in the Study; Level 2 or Above According to Functional Ambulation Classification
Keywords: Stroke; Proprioception; Lower limb functionality; Ankle joint; Balance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Humac Norm İsokinetic Machine — Tecno Body Prokin Isokinetic Balance System CSMI (CYBEX) Humac Norm Isokinetic Testing and Exercise System Romberg Test Mini Mental Test (MMSE) Fugl-Meyer Assessment of the lower limb
  Other Names: Tecno Body Prokin Isokinetic Balance System

SUMMARY:
Stroke is defined as a neurological disorder resulting from acute focal damage to the central nervous system caused by vascular factors, which may include cerebral infarction, intracerebral haemorrhage and subarachnoid haemorrhage. Postural balance is a critical factor affecting walking and gait performance in the community after stroke. Gait disorders contribute significantly to functional disability in individuals after stroke. These impairments encompass a variety of changes, including muscle weakness in the affected lower limb, resulting in reduced weight bearing on that limb. This results in a slower and less safe gait. Given the impact on gait, functional mobility is also compromised, including daily activities such as sitting, standing, walking, turning and climbing or descending stairs. Proprioception is impaired in a large percentage of individuals following stroke. The presence of proprioception deficits has been identified as an important determinant of unfavourable functional outcomes after stroke, especially in terms of achieving independence in basic activities of daily living and length of hospital stay. In the literature, there are no studies investigating the relationship between ankle position sense and lower extremity functionality with balance and falls using Humac Norm Isokinetic Machine and Tecno Body Prokin Isokinetic Balance System simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 40-80 years
* Volunteering to participate in the study

Exclusion Criteria:

* Being diagnosed with vertigo
* Having a history of serious neurological diseases such as Parkinson's disease, multiple sclerosis except hemiplegia
* Having a previous operation for the lower limb
* Poor co-operation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with haemiplegia after stroke
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Tecno Body Prokin Isokinetic Balance System | First Day
  It expresses the equilibrium rate and the probability of falling.
CSMI (CYBEX) Humac Norm Isokinetic Test and Exercise System | First day
  Measures ankle joint position sensation.
Berg Balance Scale | First day
  It was developed for the evaluation of postural dominance.
Fugl-Meyer Assessment of the lower extremity | First day
  Is used for the assessment of motor function after stroke. The total possible score for the lower limb is 34. The higher the score, the better the performance.
Tinetti Fall Activity Scale | First day
  It measures how confident the individual is in performing some activities of daily living such as reaching shelves, walking around the house, dressing and undressing, and personal care without falling. There is a rating between 1-10. Each question is defined as 1 (very confident), 10 (not confident at all). If the total score is >70, there is fear of falling.
Time Up Go Test | First day
  The purpose of the test is to provide an approach to observing gait. The patient is observed and timed while getting up from the chair, walking 3 metres, turning, walking back and sitting again.
Mini Mental Test | First day
  The MMSE (Mini-Mental State Examination) is a 30-question assessment tool commonly used by health professionals to assess cognitive functioning, including elements such as thinking, communication, comprehension and memory, to detect potential disorders.
Romberg Test | First day
  The Romberg sign is a potential indicator of a neurological disorder linked to proprioception, impairing the visual and vestibular elements that are crucial for maintaining balance.

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Demirel, Study Director — Izzet Baysal Physiotherapy and Rehabilitation Training and Research Hospital
Locations (1):
- Izzet Baysal Physical Therapy and Rehabilitation Education and Research Hospital, Bolu, Turkey (Türkiye)